CLINICAL TRIAL: NCT06551389
Title: Follow-up of the Systemic Lupus Erythematosus Cohort as Part of the Multidisciplinary Consultation at Brest CHRU
Acronym: COLUPUS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: COLUPUS (2017.CE.10)
Record Dates: First submitted 2019-06-20; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: autoimmune diseases; joint diseases; cutaneous systemic diseases; musculoskeletal diseases; arthritis; rheumatoid; rheumatic diseases; connectivite tissue diseases; immune system diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases; Joint Diseases; Musculoskeletal Diseases; Arthritis; Rheumatic Diseases; Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Biosamples in routine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Systemic lupus erythematosus is a complex systemicautoimmune disease that can affect most organs of the human body.

Although they are many recommendations on the diagnosis and managment of SLE, diagnosis and therapeutic managment is still challenging.

A pluridisciplinary consultation grouping rheumatologist, nephrologist, dermatologist, gynecologist, internist and immunologists has been set up in 2009 at the university hospital of Brest.

The investigators would like to identify in a longitudinal cohort the occurrence of the different clinico-biological and immunological patterns of systemic lupus erythematosus patients during our multidisciplinary consultation.

It is now crucial to organize a standardized data collection of these patients in order to evaluate our pratices, to be able to study the epidemiology of SLE in our city, and to promote this initiative at national and international level.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over 18 years old of the multidisciplinary consultation

Exclusion Criteria:

* Opposition of patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the systemic lupus erythematous's multidisciplinary consultation at Brest CHRU
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-01-17 (Actual); Primary Completion 2027-01-17 (Estimated); Study Completion 2027-01-17 (Estimated)

PRIMARY OUTCOMES:
Cohort data | one year
  Prevalence and incidence of the clinico-biological and immunological patterns in a longitudinal cohort present in the standardized collection book including evaluation of différents criteria aspects : SLICC criteria
Cohort data | one year
  Prevalence and incidence of the clinico-biological and immunological patterns in a longitudinal cohort present in the standardized collection book including evaluation of différents criteria aspects : SLEDAI score
Cohort data | one year
  Prevalence and incidence of the clinico-biological and immunological patterns in a longitudinal cohort present in the standardized collection book including evaluation of différents criteria aspects : SDI score

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France